CLINICAL TRIAL: NCT07290101
Title: A Prospective, Single-Center, First-in-Man Clinical Trial to Evaluate the Safety and Feasibility of the Bioresorbable Peripheral Balloon-Expandable Covered Scaffold System in Patients With Iliac Artery Stenosis or Occlusion Lesions
Brief Title: A First-in-Man Clinical Trial to Evaluate the Safety and Feasibility of ICS-Elpis in Patients With Iliac Artery Stenosis or Occlusion Lesions
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Biotyx Medical (Shenzhen) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: ICS-FIM
Record Dates: First submitted 2025-12-04; First posted 2025-12-18 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Iliac Artery Stenosis; Iliac Artery Occlusion
Keywords: iliac artery occlusion; Bioresorbable Peripheral Balloon-Expandable Covered Scaffold System; iliac artery stenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ICS-Elpis (Experimental): Bioresorbable Peripheral Balloon-Expandable Covered Scaffold System
  Interventions: Device: Bioresorbable Peripheral Balloon-Expandable Covered Scaffold System

INTERVENTIONS:
Device: Bioresorbable Peripheral Balloon-Expandable Covered Scaffold System — Subjects in the arm will be treated with ICS-Elpis

SUMMARY:
This trial is a prospective, single-center, first-in-man clinical trial to evaluate the feasibility, preliminary safety and effectiveness of the Bioresorbable Peripheral Balloon-Expandable Covered Scaffold System. 15 subjects are intended to be enrolled.

DETAILED DESCRIPTION:
Clinical follow-up visits should be conducted at before discharge, 30 days, 6 month, 9 months, and 12 months post-procedure. CTA and DUS will be performed at 6 month and 12 months post-procedure.

The primary endpoints include primary patency rate of the target lesion at 12 months post-procedure and Major Adverse Events (MAE) at 9 months post-procedure.

ELIGIBILITY:
Inclusion Criteria:

General inclusion criteria

1. Patients with stenosis or occlusion of the common iliac artery and/or external iliac artery caused by atherosclerosis.
2. Age between 18 - 85 years old. Male or non-pregnant female.
3. Patients with intermittent claudication (Rutherford category 2-3) or ischemic rest pain (Rutherford category 4).
4. Patients who can understand the purpose of the trial, voluntarily participate and sign the informed consent form, and are willing to complete the follow-up according to the protocol requirements.

Angiographic Inclusion Criteria

1. Patients with evidence of unilateral or bilateral de novo or restenosis (non-stent treatment) lesion(s) in the common iliac artery and/or external iliac artery, with the stenosis degree of the target lesion being≥50% (including occlusion).
2. The target lesion(s) can be successfully crossed with a guide wire and pre-dilated with an appropriately sized balloon.
3. The target lesion(s) with reference vessel diameter between 4.0 mm and 12.0 mm, and total length of unilateral lesion(s) ≤ 100 mm (tandem lesions are allowed).
4. Up to two ipsilateral target lesions or bilateral lesions are allowed (one target lesion per limb, with the length adhering to the unilateral criterion). Up to two stents are allowed for stent overlap per side (i.e., a maximum of two stents can be implanted per side).
5. Patients with angiographic evidence of patent outflow vessels in the target limb, including: a healthy common femoral artery (<50% stenosis); at least one of the deep femoral artery or superficial femoral artery is patent (<50% stenosis); a healthy popliteal artery (<50% stenosis); and at least one patent infrapopliteal vessel connected (<50% stenosis).
6. For stenotic or occlusive target lesion(s) located at the ostium of the common iliac artery without a residual stump, intervention can be achieved through kissing stent technique.

Exclusion Criteria:

General exclusion criteria

1. Patients with previously stented target lesion.
2. Patients who have undergone lower extremity arterial intervention within 30 days before the index procedure, or has such intervention planned for within 30 days after the index procedure.
3. Patients with a history of or planned ipsilateral aortoiliac bypass surgery during the index procedure.
4. Patients who were expected to undergo amputation of the target limb before the index procedure.
5. Patients with an aneurysm, perforation and/or dissection of the target iliac artery before the index procedure.
6. Patients who have undergone coronary artery intervention within 30 days before the index procedure, or has such intervention planned for within 30 days after the index procedure (including the index procedure).
7. Patients with acute myocardial infarction or angina pectoris within 30 days before the index procedure.
8. Patients with a stroke within 3 months before the index procedure, or a stroke more than 3 months before the index procedure accompanied by severe paralysis and aphasia sequelae.
9. Patients with known intolerance to antiplatelet, anticoagulant, or thrombolytic medications.
10. Patients with known diseases (not related to the trial) that require indefinite or lifelong anticoagulation therapy.
11. Patients with known allergies to aspirin, heparin, clopidogrel, contrast agent, poly(lactide), iron and its degradation products.
12. Patients with a history of iron overload or iron disorder, such as hereditary hemochromatosis, etc.
13. Patients with coagulation insufficiency (platelet count < 80*109/L), systemic coagulation disorders or hypercoagulable tendencies.
14. Patients with severe hepatic or renal insufficiency (serum creatinine >2 times the upper limit of normal or on renal dialysis; ALT or AST > 5 times the upper limit of normal).
15. Patients with a life expectancy of less than two years.
16. Patient currently participating in another clinical trial, and have not yet completed that trial.
17. Patients who are not suitable for participating the trial as per investigator judgement.

Angiographic Exclusion Criteria

1. Patients with angiographic evidence of thrombus within or adjacent to the target lesion(s).
2. Patients with a history of ipsilateral iliac artery stenting, where the distance between the previously implanted stent and the current target lesion is ≤ 5 mm.
3. Patients with coexisting ipsilateral iliac aneurysms or abdominal aortic aneurysms.
4. Patients in whom the internal iliac artery is patent, but implanting the stent in the target lesion will block the blood flow from entering the internal iliac artery.
5. Patients requiring placement of a study device within 2 cm proximal to the inguinal ligament.
6. Patients with severe calcification of the target lesion which makes it impossible for the pre-dilation balloon to reach its nominal diameter.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-12-08 (Estimated); Primary Completion 2027-12-01 (Estimated); Study Completion 2028-03-01 (Estimated)

PRIMARY OUTCOMES:
Primary Efficacy Endpoint: Primary Patency Rate of the Target Lesion | At12 months
  Primary patency is defined as the peak systolic velocity ratio (PSVR) ≤2.4 assessed by duplex ultrasonography (DUS) or the stenosis degree of the target lesion≤70% assessed by CTA; if there is a conflict between the results of DUS and CTA, the CTA result should prevail.
Primary Safety Endpoint: Rate of Major Adverse Events | At 30 days (for death and MI) and 9 months (for TLR and major amputation)
  The endpoint is a composite endpoint includes
  1. Device or procedure-related death within 30 days
  2. Myocardial Infarction (MI) within 30 days,
  3. Target lesion revascularization (TLR) within 9 months,
  4. Major amputation above the ankle joint of the target limb, resulting from a vascular event within 9 months.

CONTACTS AND LOCATIONS:
Locations (1):
- Renji Hospital Affiliated to Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided